CLINICAL TRIAL: NCT00080938
Title: A Phase II Study of Temozolomide and Radiation Therapy in Patients With Brain Metastasis From Non-small Cell Lung Cancer (NSCLC)
Brief Title: Temozolomide and Radiation Therapy in Treating Patients With Brain Metastasis Secondary to Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000357567; U10CA021115 (NIH); E1F03 (Other: Eastern Cooperative Oncology Group (ECOG))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; squamous cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; bronchoalveolar cell lung cancer; adenosquamous cell lung cancer; tumors metastatic to brain
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Brain Neoplasms | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide and Radiation (Experimental): Temozolomide:administered orally. Radiation: whole brain radiation therapy
  Interventions: Drug: Temozolomide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Temozolomide — Temozolomide (TMZ) to be given at a dose of 75 mg/m2/day for 14 days, starting on D1 of whole brain radiotherapy (WBRT). Three weeks after completion of WBRT, TMZ will be given at a dose of 200 mg/m2/day x 5 days (or 150 mg/m2/day if prior chemotherapy) every 28-days,for an additional two cycles.
  Other Names: Temodar
Radiation: Radiation therapy — Standard whole brain radiation therapy 30 Gy in ten fractions.
  Other Names: Whole brain radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as temozolomide may make the tumor cells more sensitive to radiation therapy. Combining temozolomide with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with whole-brain radiation therapy works in treating patients with brain metastasis secondary to non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the intracranial response rate in patients with brain metastasis secondary to non-small cell lung cancer treated with whole brain radiotherapy and temozolomide.

Secondary

* Determine the time to radiological progression in patients treated with this regimen.
* Determine the time to neurological progression (confirmed by magnetic resonance imaging (MRI)) in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo whole brain radiotherapy once daily, 5 days a week, for 2 weeks (10 fractions). Patients also receive concurrent oral temozolomide once daily on days 1-14.

Beginning 3 weeks after the completion of chemoradiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of neurologic (Central Nervous System, CNS) progression or unacceptable toxicity.

Patients were followed every 3 months for 2 years.

ACCRUAL: A total of 26 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC), including the following histologies:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell carcinoma
  * Bronchoalveolar carcinoma
  * All variants of NSCLC
* At least 1 bidimensionally measurable brain metastasis

  * Confirmed by MRI within the past two weeks, and computed tomography (CT) scan is not acceptable
  * Biopsy is not required
  * Not eligible for surgical resection or radiosurgery of brain metastasis
* Systemic disease not in immediate need of chemotherapy
* Age>=18 years
* ECOG Performance status of 0-1
* More than 12 weeks of life expectancy
* Adequate hematologic, renal, and liver function as demonstrated by laboratory values performed within two weeks, inclusive, prior to administration of study drug or registration

  * Absolute neutrophil count ≥ 1,500/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Hemoglobin ≥ 10 g/dL
  * Bilirubin ≤ 2 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2 times upper limit of normal (5 times ULN if liver metastases are present)
  * Alkaline phosphatase ≤ 2 times ULN (5 times ULN if liver metastases are present)
  * Creatinine ≤ 1.6 mg/dL
* Fertile patients must use effective contraception
* Prior biologic therapy allowed
* More than 4 weeks since prior chemotherapy
* Prior radiotherapy for local control or palliative therapy for painful bony lesions allowed
* Prior surgery for brain metastasis allowed
* At least 4 weeks since prior radiotherapy to ≥ 15% of bone marrow (2 weeks for < 15% of bone marrow) and recovered

  * No prior radiotherapy to ≥ 50% of bone marrow
* Concurrent radiotherapy to painful bony lesions allowed provided no more than 15% of bone marrow is irradiated

Exclusion Criteria:

* HIV positive
* AIDS-related illness
* Poor medical risks due to active nonmalignant systemic disease
* Frequent vomiting
* There is medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction)
* Pregnant or nursing
* Prior temozolomide
* Prior radiotherapy to the brain, including stereotactic radiosurgery to a different lesion
* Concurrent intensity modulated radiotherapy or 3-D cranial radiotherapy
* Other concurrent investigational agents
* Other concurrent treatment for brain metastasis
* Other concurrent chemotherapy during study radiotherapy
* Concurrent growth factors to induce elevations in blood counts for the purposes of administration of study drug at scheduled dosing interval or to allow treatment with study drug at a higher dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-12-20 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. I. Robins, MD, PhD, Study Chair — University of Wisconsin, Madison

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Activated on 10/18/2005, accrued its first patient on 12/20/2005, terminated on 3/13/2007. Institutes include Mayo Clinic Rochester, Northwestern University, Wisconsin, University of, Stanford University, Lankenau Hospital,Toledo Community Hosp Onc Prog CCOP,Sanford Cancer Ctr-Oncology Clinic,Carle Cancer Center CCOP
Groups:
- Temozolamide and Radiation: Patients were to receive whole brain radiation therapy (WBRT), 30 Gy in ten fractions, plus Temozolomide (TMZ) given at a dose of 75 mg/m2/day for 14 days starting on day 1 of radiotherapy. Three weeks after completion of WBRT, TMZ was to be given at a dose of 200 mg/m2/day x 5 days (or 150 mg/m2/day if prior chemotherapy) every 28 days for up to 6 cycles post WBRT (for a total of 7 cycles of protocol treatment).
Period: Overall Study
Arm/Group | Temozolamide and Radiation
Started | 26
Began Protocol Therapy | 25
Eligible and Treated | 21
Completed | 2
Not Completed | 24
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 6
Not completed — Death | 2
Not completed — Lack of Efficacy | 7
Not completed — other disease | 1
Not completed — Not started protocol therapy | 1
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Arm/Group | Temozolamide and Radiation
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Intracranial Response
Description: Response was assessed per Response Evaluation Criteria in Solid Tumor (RECIST) by brain MRI in the 21 eligible and treated patients.Complete response (CR): complete disappearance of the clinically detectable malignant brain metastasis(es) being followed on MRI scan off corticosteroids and a stable or improving neurologic exam. Partial response (PR): greater than or equal to a 50% reduction in the sum of the product(s) of the maximal cross-sections on MRI scan with a stable or decreasing dose of corticosteroids and a stable or improving neurologic exam. Response = CR + PR
Time Frame: assessed every cycle while on treatment, then every 3 months for 2 years
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | Temozolamide and Radiation
Number analyzed (Participants) | 21
participants | 3

2. Secondary Outcome: 1-year Neurologic (Central Nervous System, CNS) Progression Free Rate
Description: 1-year CNS progression free rate is the percentage of patients who had no CNS progression after being followed for 1 year . Progressive disease (CNS) was defined as a 25% or greater increase in the sum of the product(s) of the maximal cross-sections on MRI scan, reappearance of any lesion that has disappeared, development of any new lesion(s), stable disease with a deterioration of neurologic exam, or clear worsening of any evaluable disease.
Time Frame: assessed every 3 months for 2 years
Population: Eligible, treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Temozolamide and Radiation
Number analyzed (Participants) | 21
percentage of participants | 90.5 [69.6 to 98.8]

3. Secondary Outcome: Time to Non-CNS (Systemic) Progression
Description: Time to non-CNS progression was calculated from time of protocol entry to time of first systemic progressive disease or death. Patients alive and non-CNS progression-free at last follow-up were censored. Disease progression was defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter (per RECIST criteria). Development of new lesions in non-CNS sites also constituted non-CNS progression. The 21 eligible and treated patients were included in the analysis.
Time Frame: assessed every 3 months for 2 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolamide and Radiation
Number analyzed (Participants) | 21
months | 3.2 [1.3 to 5.7]

4. Secondary Outcome: Overall Survival Time
Description: Overall survival (months) was calculated from time of protocol entry to time of death from any cause. Patients alive at last follow-up were censored. The 21 eligible and treated patients were included in the analysis.
Time Frame: assessed every 3 months for 2 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolamide and Radiation
Number analyzed (Participants) | 21
months | 7 [3.9 to 16.6]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (cycle 1=35 days, All other cycles =28 days) while on treatment and for 30 days after the end of the treatment
Arm/Group | Temozolamide and Radiation
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolamide and Radiation (N=25)
Anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Investigations) | 1
Fatigue (General disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Muco/stomatitis by exam,oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Infection Gr0-2 neut, blood (Infections and infestations) | 1
CNS, hemorrhage (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Temozolamide and Radiation (N=25)
Anemia (Blood and lymphatic system disorders) | 11
Leukopenia (Investigations) | 4
Thrombocytopenia (Investigations) | 8
Fatigue (General disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 9
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Radiation dermatitis (Injury, poisoning and procedural complications) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Muco/stomatitis by exam,oral cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Taste disturbance (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
ALT Increased (Hepatobiliary disorders) | 6
AST Increased (Hepatobiliary disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No